CLINICAL TRIAL: NCT01597687
Title: Bordetella Pertussis Infection Among Adolescents and Adults With Prolonged Cough
Brief Title: Pertussis Infection in Adolescents and Adults With Prolonged Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 115741
Record Dates: First submitted 2012-05-03; First posted 2012-05-14 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-06

CONDITIONS: Pertussis
Keywords: pertussis infection; Prevalence; health economic burden; prolonged cough
MeSH Terms: conditions — Whooping Cough | interventions — Blood Specimen Collection; Data Collection

ARMS (3):
- Malaysia Group (Experimental): Malaysian adults aged >19 years with prolonged cough of 2 weeks or more.
  Interventions: Procedure: Blood collection; Other: Data collection
- Taiwan Group (Experimental): Taiwanese adults aged >19 years with prolonged cough of 2 weeks or more.
  Interventions: Procedure: Blood collection; Other: Data collection
- Thailand Group (Experimental): Thailandese adults aged >19 years with prolonged cough of 2 weeks or more.
  Interventions: Procedure: Blood collection; Other: Data collection

INTERVENTIONS:
Procedure: Blood collection — 1 blood sample will be collected from each subject.
Other: Data collection — Quality of Life and HE questionnaires.

SUMMARY:
This study aims to determine the burden of pertussis infection among adolescents and adults with prolonged cough in four Asian countries, namely Malaysia, Philippines, Taiwan and Thailand. This study also aims to assess the health economic (HE) impact of pertussis.

DETAILED DESCRIPTION:
Data from this cross-sectional study will be useful in reviewing the need for introduction of booster doses of pertussis vaccines in adolescent and adult population in Malaysia, Philippines, Taiwan and Thailand.

This study will enrol patients with prolonged cough of 2 weeks or more and detect pertussis with serological tests in order to estimate the prevalence of pertussis infection among such patients. No vaccine will be administered during this study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13-18 years or adults aged >18years.
* Presenting with prolonged cough of 2 weeks (14 days) or more.
* Subjects who the investigator believes that they/ their parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject/ from the parent(s)/LAR of the subject. If the subject below the age of consent is legally eligible, his/her signature on the informed assent form should be obtained.

Exclusion Criteria:

* Child in care.
* Subjects with known chronic cough-causing disease and immunodeficiency.
* Subjects treated with angiotensin-converting enzyme inhibitors (ACEI), within the past 4 weeks (28 days).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2013-05-02 (Actual); Study Completion 2013-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Malaysia (2):
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Seremban
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taoyuan District
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Songkhla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koh MT, Liu CS, Chiu CH, Boonsawat W, Watanaveeradej V, Abdullah N, Zhang X, Devadiga R, Chen J. Under-recognized pertussis in adults from Asian countries: a cross-sectional seroprevalence study in Malaysia, Taiwan and Thailand. Epidemiol Infect. 2016 Apr;144(6):1192-200. doi: 10.1017/S0950268815002393. Epub 2015 Oct 15. PMID 26468043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The duration of enrolment of all subjects was less than a year. Each subject attended one study visit at the time of enrolment, during which Quality of Life (QoL) and Health Economics (HE) questionnaires were administered and one blood sample was drawn.
Pre-assignment Details: A total of 337 subjects were enrolled into this study, but only 312 had valid laboratory results. 2 subjects were excluded due to vulnerable conditions, 16 subjects were excluded due to protocol violation and 7 subjects were excluded due to vaccination with pertussis vaccines within 1 year before blood sample collection.
Period: Overall Study
Arm/Group | Malaysia Group | Taiwan Group | Thailand Group
Started | 76 | 89 | 147
Completed | 76 | 89 | 147
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Malaysia Group | Taiwan Group | Thailand Group | Total
Number analyzed (Participants) | 76 | 89 | 147 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.08 (16.76) | 39.20 (12.29) | 42.66 (15.73) | 42.99 (15.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 60 | 101 | 210
  Male | 27 | 29 | 46 | 102
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Serological Evidence of Pertussis Infection
Description: Serological evidence of pertussis infection was defined as anti-pertussis toxin (PT) immunoglobulin G (IgG) level indicative of active or recent infection. The parameters presented were defined as follows: Seropositive = Subjects with anti-PT IgG ELISA levels ≥10 IU/ml , Seronegative = Subjects with anti-PT IgG ELISA levels < 10 IU/ml , Sero-confirmed infection = Subjects with anti-PT IgG ELISA levels ≥62.5 IU/ml , Active infection 1= Anti-PT IgG ELISA levels ≥ 100 IU/ml indicative of active or recent infection, Active infection 2 = Anti-PT IgG ELISA levels ≥ 125 IU/ml indicative of active or recent infection
Time Frame: At time of blood sampling (Day 0)
Population: The analysis was done on the According-to-Protocol (ATP) cohort which included all subjects with valid laboratory results.
Measure: Count of Participants; unit: Participants
Arm/Group | Malaysia Group | Taiwan Group | Thailand Group
Number analyzed (Participants) | 76 | 89 | 147
Participants
  Seronegative | 50 | 74 | 84
  Seropositive | 26 | 15 | 63
  Sero-confirmed infection | 6 | 1 | 9
  Active infection 1 | 1 | 0 | 3
  Active infection 2 | 0 | 0 | 2

2. Secondary Outcome: Number of Participants With Specific Clinical Features
Description: Clinical features assessed included paroxysm, whoop, night cough, cyanosis, fever post-tussive vomiting, apnoea, cyanosis, coughing up phlegm, sneezes, wheezes, episodes of being unable to stop coughing and breathlessness/chest pain.
Time Frame: At time of clinical data collection prior to enrolment (Day 0)
Population: The analysis was done on the ATP cohort for immunogenicity which included all subjects with valid laboratory results. For this outcome the subjects were grouped by their infection status: Subjects with Sero-confirmed infection and Subjects with Non-sero-confirmed infection.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Sero-confirmed Infection: Adults aged >19 years with prolonged cough of 2 weeks or more, with with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml.
- Subjects With Non-sero-confirmed Infection: Adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels < 62.5 IU/m
Arm/Group | Subjects With Sero-confirmed Infection | Subjects With Non-sero-confirmed Infection
Number analyzed (Participants) | 16 | 296
Participants
  Whoop: Yes | 2 | 18
  Whoop: No | 14 | 278
  Paroxysm: Yes | 12 | 143
  Paroxysm: No | 4 | 153
  Post tussive vomiting: Yes | 6 | 72
  Post tussive vomiting: No | 10 | 224
  Apnoea: Yes | 0 | 3
  Apnoea: No | 16 | 293
  Cyanosis: Yes | 0 | 0
  Cyanosis: No | 16 | 296
  Coughing up phlegm: Yes | 6 | 180
  Coughing up phlegm: No | 10 | 116
  Sneezes: Yes | 6 | 111
  Sneezes: No | 10 | 185
  Wheezes: Yes | 3 | 34
  Wheezes: No | 13 | 262
  Cough at night: Yes | 11 | 211
  Cough at night: No | 5 | 85
  Episodes of being unable to stop coughing: Yes | 7 | 140
  Episodes of being unable to stop coughing: No | 9 | 156
  Breathlessness /chest pain: Yes | 10 | 106
  Breathlessness /chest pain: No | 6 | 190

3. Secondary Outcome: Assessment of Health Economical Impact - Number of Days Absent From Work Due to Cough
Description: Absenteeism was assessed as the mean number of days missed from work due to cough.
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥ 62.5 IU/ml, and with available data.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Malaysian Sero-confirmed Subjects Group: Malaysian adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
- Taiwanese Sero-confirmed Subjects Group: Taiwanese adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
- Thailandese Sero-confirmed Subjects Group: Thailandese adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 4 | 1 | 9
Days
  Number of days absent from work due to cough | 7.75 (14.84) | 0.00 (NA) — No absences from work due to cough were reported, hence Standard Deviation cannot be computed. | 0.22 (0.67)
  Number of paid leave days due to cough | 0.25 (0.50) | 0.00 (NA) — No absences from work due to cough were reported, hence Standard Deviation cannot be computed. | 0.22 (0.67)
  Number of unpaid leave days due to cough | 7.50 (15.00) | 0.00 (NA) — No absences from work due to cough were reported, hence Standard Deviation cannot be computed. | 0.00 (NA) — No unpaid leave days due to cough were reported, hence Standard Deviation cannot be computed.

4. Secondary Outcome: Assessment of Health Economical Impact - Number of Sero-confirmed Subjects With Loss of Income Due to Missing Work
Description: Loss of income due to missing work for sero-confirmed subjects was measured in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM), Taiwan - New Taiwan dollar (NTD), Thailand - Thai baht (BAHT).
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
Measure: Count of Participants; unit: Participants
Groups:
- Malaysia Sero-confirmed Subjects Group: Malaysian adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml.
- Taiwan Sero-confirmed Subjects Group: Taiwanese adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml.
- Thailand Sero-confirmed Subjects Group: Thailandese adults aged >19 years with prolonged cough of 2 weeks or more, with anti-pertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml.
Arm/Group | Malaysia Sero-confirmed Subjects Group | Taiwan Sero-confirmed Subjects Group | Thailand Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 1 | 9
Participants
  Loss of income due to missing work: Yes | 1 | 0 | 0
  Loss of income due to missing work: No | 3 | 1 | 9
  Loss of income due to missing work: Unknown/Not applicable | 2 | 0 | 0
  Average income loss/day >300 local currency units: Yes | 1 | 0 | 0
  Average income loss/day >300 local currency units: No | 0 | 0 | 0
  Average income loss/day >300 local currency units: Unknown/Not applicable | 5 | 1 | 9

5. Secondary Outcome: Assessment of Health Economical Impact - Number of Visits to Specific Healthcare Resources
Description: Healthcare resource utilization was assessed by the mean number of visits to any type of physicians.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Visits to physician
Arm/Group | Malaysia Sero-confirmed Subjects Group | Taiwan Sero-confirmed Subjects Group | Thailand Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 1 | 9
Visits to physician
  Number of visits to GP/ family physician clinic | 3.17 (2.40) | 0.00 (NA) — No visits to GP/ family physician clinic were reported, hence Standard Deviation could not be computed. | 1.00 (1.00)
  Number of visits to Specialist clinic | 0.33 (0.52) | 8.00 (NA) — Only one participant reported visits to Specialist clinic. Standard Deviation cannot be computed on a single value. | 1.00 (0.50)
  Number of visits to the Emergency room | 0.50 (0.84) | 1.00 (NA) — Only one participant reported visits to the Emergency Room. Standard Deviation cannot be computed on a single value. | 0.00 (NA) — No visits to the Emergency Room were reported, hence Standard Deviation could not be computed.
  Total healthcare visits | 4.00 (3.03) | 9.00 (NA) — Only one participant reported healthcare visits. Standard Deviation cannot be computed on a single value. | 2.00 (1.12)

6. Secondary Outcome: Assessment of Health Economical Impact - Summary of Travel Costs for Sero-confirmed Subjects - Malaysia
Description: The travel costs were assessed in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM).
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the Malaysian subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
Measure: Mean (Standard Deviation); unit: Malaysian ringgit (RM)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 0 | 0
Malaysian ringgit (RM)
  Amount for travel to consultation with GP(s) | 43.83 (54.77) |  |
  Amount for travel to consultation with specialist | 2.50 (4.18) |  |
  Amount for travel to Emergency room(s) | 9.17 (16.25) |  |
  Total cost for transportation | 55.50 (63.71) |  |

7. Secondary Outcome: Assessment of Health Economical Impact - Summary of Travel Costs for Sero-confirmed Subjects - Taiwan
Description: The travel costs were assessed in the local currency of each country, as follows: Taiwan - New Taiwan dollar (NTD)
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the Taiwanese subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
Measure: Mean (Standard Deviation); unit: New Taiwan dollar (NTD)
Groups:
- Malaysian Sero-confirmed Subjects Group: Malaysian adults aged >19 years with prolonged cough of 2 weeks or more, with antipertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
- Taiwanese Sero-confirmed Subjects Group: Taiwanese adults aged >19 years with prolonged cough of 2 weeks or more, with antipertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
- Thailandese Sero-confirmed Subjects Group: Thailandese adults aged >19 years with prolonged cough of 2 weeks or more, with antipertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 1 | 0
New Taiwan dollar (NTD)
  Amount for travel to consultation with GP(s) |  | 0.00 (NA) — No visits to GP/ family physician clinic were reported, hence Standard Deviation could not be computed. |
  Amount for travel to consultation with specialist |  | 2400.00 (NA) — Only one participant reported visits to Specialist clinic. Standard Deviation cannot be computed on a single value. |
  Amount for travel to Emergency room(s) |  | 300.00 (NA) — Only one participant reported visits to the Emergency Room. Standard Deviation cannot be computed on a single value. |
  Total cost for transportation |  | 2700.00 (NA) — Only one participant reported healthcare visits. Standard Deviation cannot be computed on a single value. |

8. Secondary Outcome: Assessment of Health Economical Impact - Summary of Travel Costs for Sero-confirmed Subjects - Thailand
Description: The travel costs were assessed in the local currency of each country, as follows: Thailand - Thai baht (BAHT).
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the Tailandese subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
Measure: Mean (Standard Deviation); unit: Thai baht (BAHT)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 0 | 9
Thai baht (BAHT)
  Amount for travel to consultation with GP(s) |  |  | 1133.30 (1450.90)
  Amount for travel to consultation with specialist |  |  | 668.89 (709.09)
  Amount for travel to Emergency room(s) |  |  | 0.00 (NA) — No visits to the Emergency Room were reported, hence Standard Deviation could not be computed.
  Total cost for transportation |  |  | 1802.20 (1819.20)

9. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting the GP(s) - Malaysia
Description: The medical costs were assessed in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the GP(s).
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the Malaysian subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
  One subject who reported 'out of pocket expenses' did not report 'Total medical cost'.
Measure: Mean (Standard Deviation); unit: Malaysian ringgit (RM)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 0 | 0
Malaysian ringgit (RM)
  Out of Pocket expense: number analyzed (Participants) | 4 | 0 | 0
  Out of Pocket expense | 47.50 (9.57) |  |
  Total medical cost: number analyzed (Participants) | 3 | 0 | 0
  Total medical cost | 43.33 (5.77) |  |

10. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting the GP(s) - Taiwan
Description: The medical costs were assessed in the local currency of each country, as follows: Taiwan - New Taiwan dollar (NTD). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the GP(s).
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: New Taiwan dollar (NTD)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 1 | 0
New Taiwan dollar (NTD)
  Out of Pocket expense |  | 0.00 (NA) — No visits to GP/ family physician clinic were reported, hence Standard Deviation could not be computed. |
  Total medical cost |  | 0.00 (NA) — No visits to GP/ family physician clinic were reported, hence Standard Deviation could not be computed. |

11. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting the GP(s) - Thailand
Description: The medical costs were assessed in the local currency of each country, as follows: Thailand - Thai baht (BAHT). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the GP(s).
Time Frame: At time of questionnaire administration (Day 0)
Population: The assessment was performed only on the Thailandese subjects with sero-confirmed infection, i.e with Immunoglobulin G ELISA levels ≥62.5 IU/ml, and with available data.
Measure: Mean (Standard Deviation); unit: Thai baht (BAHT)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 0 | 9
Thai baht (BAHT)
  Out of Pocket expense: number analyzed (Participants) | 0 | 0 | 7
  Out of Pocket expense |  |  | 1114.30 (1665.80)
  Total medical cost: number analyzed (Participants) | 0 | 0 | 7
  Total medical cost |  |  | 1114.30 (1665.80)

12. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Specialist Clinics - Malaysia
Description: The medical costs were assessed in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the specialist clinics.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Malaysian ringgit (RM)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 0 | 0
Malaysian ringgit (RM)
  Out of Pocket expense: number analyzed (Participants) | 4 | 0 | 0
  Out of Pocket expense | 0.00 (NA) — None of the participants with available data reported any expenses for visits to specialist clinics, hence Standard Deviation could not be computed. |  |
  Total medical cost: number analyzed (Participants) | 4 | 0 | 0
  Total medical cost | 0.00 (NA) — None of the participants with available data reported any expenses for visits to specialist clinics, hence Standard Deviation could not be computed. |  |

13. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Specialist Clinics - Taiwan
Description: The medical costs were assessed in the local currency of each country, as follows: Taiwan - New Taiwan dollar (NTD). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the specialist clinics.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: New Taiwan dollar (NTD)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 1 | 0
New Taiwan dollar (NTD)
  Out of Pocket expense |  | 1700.00 (NA) — Only one participant reported expenses for visiting specialist clinics. Standard Deviation cannot be computed on a single value. |
  Total medical cost |  | 1700.00 (NA) — Only one participant reported expenses for visiting specialist clinics. Standard Deviation cannot be computed on a single value. |

14. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Specialist Clinics - Thailand
Description: The medical costs were assessed in the local currency of each country, as follows: Thailand - Thai baht (BAHT). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the specialist clinics.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Thai baht (BAHT)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 0 | 9
Thai baht (BAHT)
  Out of Pocket expense: number analyzed (Participants) | 0 | 0 | 7
  Out of Pocket expense |  |  | 645.71 (711.87)
  Total medical cost: number analyzed (Participants) | 0 | 0 | 7
  Total medical cost |  |  | 645.71 (711.87)

15. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Emergency Rooms - Malaysia
Description: The medical costs were assessed in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the emergency rooms.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Malaysian ringgit (RM)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 0 | 0
Malaysian ringgit (RM)
  Out of Pocket expense: number analyzed (Participants) | 4 | 0 | 0
  Out of Pocket expense | 0.00 (NA) — None of the participants with available data reported any expenses for Emergency Room visits, hence Standard Deviation could not be computed. |  |
  Total medical cost: number analyzed (Participants) | 4 | 0 | 0
  Total medical cost | 0.00 (NA) — None of the participants with available data reported any expenses for Emergency Room visits, hence Standard Deviation could not be computed. |  |

16. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Emergency Rooms - Taiwan
Description: The medical costs were assessed in the local currency of each country, as follows: Taiwan - New Taiwan dollar (NTD). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the emergency rooms.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: New Taiwan dollar (NTD)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 1 | 0
New Taiwan dollar (NTD)
  Out of Pocket expense |  | 750.00 (NA) — Only one participant reported any expenses for Emergency Room visits. Standard Deviation cannot be computed for a single value. |
  Total medical cost |  | 750.00 (NA) — Only one participant reported any expenses for Emergency Room visits. Standard Deviation cannot be computed for a single value. |

17. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Emergency Rooms - Thailand
Description: The medical costs were assessed in the local currency of each country, as follows: Thailand - Thai baht (BAHT). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the emergency rooms.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Thai baht (BAHT)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 0 | 9
Thai baht (BAHT)
  Out of Pocket expense: number analyzed (Participants) | 0 | 0 | 7
  Out of Pocket expense |  |  | 0.00 (NA) — No Emergency Room visits were reported, hence Standard Deviation could not be computed.
  Total medical cost: number analyzed (Participants) | 0 | 0 | 7
  Total medical cost |  |  | 0.00 (NA) — No Emergency Room visits were reported, hence Standard Deviation could not be computed.

18. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Healthcare Resources in General - Malaysia
Description: The medical costs were assessed in the local currency of each country, as follows: Malaysia - Malaysian ringgit (RM). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the healthcare resources in general
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Malaysia - Malaysian ringgit (RM)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 0 | 0
Malaysia - Malaysian ringgit (RM)
  Out of Pocket expense: number analyzed (Participants) | 4 | 0 | 0
  Out of Pocket expense | 47.50 (9.57) |  |
  Total medical cost: number analyzed (Participants) | 3 | 0 | 0
  Total medical cost | 43.33 (5.77) |  |

19. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Healthcare Resources in General - Taiwan
Description: The medical costs were assessed in the local currency of each country, as follows: Taiwan - New Taiwan dollar (NTD). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the healthcare resources in general
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: New Taiwan dollar (NTD)
Groups:
- Thailandese Sero-confirmed Subjects Group: Thailandese adul ts aged >19 years with prolonged cough of 2 weeks or more, with antipertussis Immunoglobulin G ELISA levels ≥62.5 IU/ml
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 1 | 0
New Taiwan dollar (NTD)
  Out of Pocket expense |  | 2450.00 (NA) — Only one participant reported any expenses for visiting healthcare resources. Standard Deviation cannot be computed on a single value. |
  Total medical cost |  | 2450.00 (NA) — Only one participant reported any expenses for visiting healthcare resources. Standard Deviation cannot be computed on a single value. |

20. Secondary Outcome: Assessment of Health Economical Impact - Summary of Medical Costs for Sero-confirmed Subjects Visiting Healthcare Resources in General - Thailand
Description: The medical costs were assessed in the local currency of each country, as follows: Thailand - Thai baht (BAHT). Total medical cost included the cost spent for consultation, medicines, laboratory tests etc., for visiting the healthcare resources in general
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Thai baht (BAHT)
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 0 | 0 | 9
Thai baht (BAHT)
  Out of Pocket expense: number analyzed (Participants) | 0 | 0 | 7
  Out of Pocket expense |  |  | 1760.00 (1978.00)
  Total medical cost: number analyzed (Participants) | 0 | 0 | 7
  Total medical cost |  |  | 1760.00 (1978.00)

21. Secondary Outcome: Assessment of Health Economical Impact - Summary of Total Amount of Time Spent by Sero-confirmed Subjects Visiting Healthcare Resources in General
Description: Total amount of time spent on seeing the doctor(s) which includes the return trip and the overall time spent at clinic(s)/hospital(s) for waiting, consultation, tests, pharmacy etc.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 1 | 9
Hours
  Time spent for consultation with the GP(s) | 6.38 (8.74) | 0.00 (NA) — No consultations with the GP were reported, hence Standard Deviation could not be computed. | 2.28 (2.97)
  Time spent for consultation with the specialist(s) | 0.33 (0.52) | 20.00 (NA) — Only one participant reported any consultation with the Specialist. Standard Deviation cannot be computed on a single value. | 2.97 (3.13)
  Time spent for treatment in the emergency room(s) | 1.17 (1.83) | 3.00 (NA) — Only one participant reported time spent at the Emergency Room. Standard Deviation cannot be computed on a single value. | 0.00 (NA) — No Emergency Room visitis were reported, hence Standard Deviation could not be computed.
  Total time spent to visit the healthcare resources | 7.88 (10.52) | 23.00 (NA) — Only one participant reported time spent at any healthcare resources. Standard Deviation cannot be computed on a single value. | 5.25 (4.88)

22. Secondary Outcome: Assessment of the Impact of Pertussis on Quality of Life of Patients: Number of Participants Reporting Problems With Specific Characteristics
Description: Health-related quality of life of pertussis patients was assessed using the EQ-5D Questionnaire. The EQ-5D is composed of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), with 3 levels of severity within each dimension. The EQ-5D levels were further dichotomised into "no problems" (level 1) and "with problems" (level 2 & 3). The number of participants within these 2 levels are reported.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 1 | 9
Participants
  Mobility: No problems | 6 | 1 | 7
  Mobility: With problems | 0 | 0 | 2
  Self-Care: No problems | 6 | 1 | 9
  Self-Care: With problems | 0 | 0 | 0
  Usual Activities: No problems | 4 | 0 | 6
  Usual Activities: With problems | 2 | 1 | 3
  Pain/Discomfort: No problems | 4 | 0 | 6
  Pain/Discomfort: With problems | 2 | 1 | 3
  Anxiety/Depression: No problems | 3 | 0 | 6
  Anxiety/Depression: With problems | 3 | 1 | 3

23. Secondary Outcome: Assessment of the Impact of Pertussis on Quality of Life of Patients: Average EQ-5D Index Score
Description: Health-related quality of life of pertussis patients was assessed using the EQ-5D Questionnaire. The EQ-5D is composed of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), with 3 levels of severity within each dimension. Average of EQ-5D index score (ranging from 0 to 1; 0 being death and 1 being in perfect health) across sero-confirmed participants was reported.
Time Frame: At time of questionnaire administration (Day 0)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Malaysian Sero-confirmed Subjects Group | Taiwanese Sero-confirmed Subjects Group | Thailandese Sero-confirmed Subjects Group
Number analyzed (Participants) | 6 | 1 | 9
Scores on a scale | 0.84 (0.18) | 0.66 (NA) — Standard Deviation cannot be computed for a single value. | 0.75 (0.21)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected during the entire study period (at Day 0 from enrolment till completion of all study procedures).
Description: Only Serious Adverse Events were monitored in this trial, Other (non-serious) Adverse Events were not collected as planned per protocol.
Arm/Group | Malaysia Group | Taiwan Group | Thailand Group
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/89 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/89 | 0/147
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.